CLINICAL TRIAL: NCT05463159
Title: Effects of Transcutaneous Electrical Nerve Stimulation on Spasticity in Children With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0708
Record Dates: First submitted 2022-06-20; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): participants in this group will be given with TENS to spastic Hams, Adductor and TA along with stretchings and ROM as baseline treatment
  Interventions: Other: Transcutaneous electrical nerve stimulation
- Group B (Active Comparator): participants in this group will be given with TENS to opposite of spastic muscles, i.e. quards, abductor and dorsiflexors along with stretchings and ROM as baseline treatment
  Interventions: Other: Transcutaneous electrical nerve stimulation
- Group C (Active Comparator): participants in this group will be given with TENS to both spastic muscles and opposite of spastic muscle along with stretchings and ROM as baseline treatment
  Interventions: Other: Transcutaneous electrical nerve stimulation
- Group D (Active Comparator): participants in this group will be given with stretchings and ROM as baseline treatment
  Interventions: Other: Transcutaneous electrical nerve stimulation

INTERVENTIONS:
Other: Transcutaneous electrical nerve stimulation — All children received 30 min of conventional TENS (continuous stimulation with all parameters constant) with a frequency of 100 Hz and a pulse width of 200 µs.

SUMMARY:
Cerebral Palsy (CP) is a group of mental disorder that disrupts the person's ability of moving, maintaining their balance and posture. Cerebral palsy is a motor disorganization in Childhood. Cerebral palsy can occur before birth, during birth, within a month after birth, or during 1st year of life when brain is under development. Symptoms vary from person to person in case of severe CP child must needs the equipment used to enhance their mobility and to train muscles. Transcutaneous electrical nerve stimulation (TENS) is method of relieving pain by using mild electric current. Purpose of this study will be to determine effects of TENS on spasticity and gross motor function in children with cerebral palsy. TENS is a small machine operated with battery containing attached sticky pads known as electrodes placed on stiffed and painful area of muscles. Classified by Ashworth Scale and Modified Tardieu Scale. Subjects will be randomly divided into four groups 1) Group A= TENS on spastic muscle/agonist, 2) Group B= TENS on antagonist, 3) GroupC= TENS on both agonist and antagonist muscle, Group D= conventional physiotherapy total treatment period is about 3 to 6 weeks. This study will help to discuss how much extent TENS will effect spasticity in children with cerebral palsy. Data will be analyzed through SPSS 22

ELIGIBILITY:
Inclusion Criteria:

* Age 6-12
* Both Male and Female
* Spastic Cerebral Palsy

Exclusion Criteria:

* Patients with History of uncontrolled seizures
* Patients undergoing previous tendon lengthening surgery
* History of Botox Injection

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-08-15 (Estimated)

PRIMARY OUTCOMES:
Change in Modified Ashworth Scale | Baseline and 4th week
  The modified Ashworth scale(MAS) is a 6-point rating scale that is used to measure muscle tone.
  0 No increase in tone
  1 slight increase in tone giving a catch when slight increase in muscle tone, manifested by the limb was moved in flexion or extension.
  1+ slight increase in muscle tone, manifested by a catch followed by minimal resistance throughout (ROM ) 2 more marked increase in tone but more marked increased in muscle tone through most limb easily flexed 3 considerable increase in tone, passive movement difficult 4 limb rigid in flexion or extension
Change in Modified Tardieu Scale | Baseline and 4th week
  The Modified Tardieu Scale (MTS) is an often-recommended spasticity assessment.The MTS classifies the response of a relaxed muscle to a fast, passive stretch (V3). The assessment protocol involves a clinician moving the joint "as fast as possible" through its full range of motion (ROM) without specifying or measuring the speed of completion. The MTS is applied according to this standardized protocol regardless of the functional status or goals of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Fareeha Kausar, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- DHQ Hospital, Vehari, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alhusaini AA, Fallatah S, Melam GR, Buragadda S. Efficacy of transcutaneous electrical nerve stimulation combined with therapeutic exercise on hand function in children with hemiplegic cerebral palsy. Somatosens Mot Res. 2019 Mar;36(1):49-55. doi: 10.1080/08990220.2019.1584555. Epub 2019 Mar 26. PMID 30913943
- [Background] Solopova IA, Sukhotina IA, Zhvansky DS, Ikoeva GA, Vissarionov SV, Baindurashvili AG, Edgerton VR, Gerasimenko YP, Moshonkina TR. Effects of spinal cord stimulation on motor functions in children with cerebral palsy. Neurosci Lett. 2017 Feb 3;639:192-198. doi: 10.1016/j.neulet.2017.01.003. Epub 2017 Jan 4. PMID 28063935
- [Background] Bakaniene I, Urbonaviciene G, Janaviciute K, Prasauskiene A. Effects of the Inerventions method on gross motor function in children with spastic cerebral palsy. Neurol Neurochir Pol. 2018 Sep-Oct;52(5):581-586. doi: 10.1016/j.pjnns.2018.07.003. Epub 2018 Jul 20. PMID 30061001
- [Background] Alabdulwahab SS. Electrical stimulation improves gait in children with spastic diplegic cerebral palsy. NeuroRehabilitation. 2011;29(1):37-43. doi: 10.3233/NRE-2011-0675. PMID 21876294
- [Background] Alabdulwahab SS, Al-Gabbani M. Transcutaneous electrical nerve stimulation of hip adductors improves gait parameters of children with spastic diplegic cerebral palsy. NeuroRehabilitation. 2010;26(2):115-22. doi: 10.3233/NRE-2010-0542. PMID 20203376